CLINICAL TRIAL: NCT01536951
Title: A Placebo-Controlled, Single Dose, Dose Escalation (Part A) and a Placebo- and Positive-Controlled Study of the Effect on the Electrocardiographic QT Interval of a Single Dose (Part B) of LY3009104 in Healthy Subjects
Brief Title: A Study of LY3009104 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14448; I4V-MC-JADO (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Healthy Participants
MeSH Terms: interventions — baricitinib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo matching LY3009104 tablets in size and appearance will be administered orally in 1 out of 3 study periods in Part A and Part B.
  Interventions: Drug: Placebo
- LY3009104 (Experimental): Part A. Single escalating dose of up to 40 milligrams (mg) of LY3009104 administered orally in 2 out of 3 study periods separated by at least a 3 day wash-out period between each dose.
  Part B. Single dose of LY3009104 determined in Part A administered orally in 1 out of 3 study periods separated by at least a 3 day wash-out period between each period.
  Interventions: Drug: LY3009104
- 400 mg moxifloxacin (Active Comparator): Part B. 400 mg moxifloxacin will be administered orally in 1 out of 3 study periods separated by at least a 3 day wash-out period between each period.
  Interventions: Drug: moxifloxacin

INTERVENTIONS:
Drug: LY3009104 — administered orally
  Other Names: Baricitinib
  Arms: LY3009104
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: moxifloxacin — Administered orally
  Arms: 400 mg moxifloxacin

SUMMARY:
This will be a 2-part, randomized, participant- and investigator-blind study in healthy males and females.

Part A of this study is to determine a safe and tolerable single oral dose of LY3009104 that yields drug exposures slightly exceeding typical exposures anticipated from repeated administration of an efficacious dose to participants. The concentration of the drug in the blood stream will be measured and information about any side effects that may occur will also be collected.

Part B of this study is to evaluate the effect of LY3009104 on the electrical activity of the heart as measured by electrocardiogram (ECG) in relation to placebo following a single oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females as determined by medical history and physical examination. Are drug free, disease free, and no cardiac abnormalities.
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have a clinically normal screening ECG with a measurable QT interval as judged by the investigator, and which in Part B allows accurate measurements of QT interval.

Exclusion Criteria:

* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participating in the study or affects or confounds the corrected QT (QTc) analysis or have QTc greater than 450 milliseconds (msec).
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had 2 parts. Part A: single-dose, dose-escalating study of LY3009104 [up to 40 milligrams (mg)] or placebo administered in each period. Part B: assessed the electrophysiological effects of a single supratherapeutic LY3009104 dose compared to a positive control (moxifloxacin) and placebo. Participants enrolled in either Part A or Part B.
Groups:
- Part A: Placebo, 30 mg LY3009104, 40 mg LY3009104: First Intervention: Placebo tablets [matching 20-mg LY3009104] administered orally once.
  Second Intervention: 30-mg LY3009104 dose administered orally once.
  Third Intervention: 40-mg LY3009104 dose administered orally once.
  There was a washout of at least 3 days between each intervention.
- Part A: 20 mg LY3009104, 30 mg LY3009104, Placebo: First Intervention: 20-mg LY3009104 dose administered orally once.
  Second Intervention: 30-mg LY3009104 dose administered orally once.
  Third Intervention: Placebo tablets (matching 40-mg LY3009104) administered orally once.
  There was a washout of at least 3 days between each intervention.
- Part A: 20 mg LY3009104, Placebo, 40 mg LY3009104: First Intervention: 20-mg LY3009104 dose administered orally once.
  Second Intervention: Placebo tablets (matching 30-mg LY3009104) administered orally once.
  Third Intervention: 40-mg LY3009104 dose administered orally once.
  There was a washout of at least 3 days between each intervention.
- Part B: 40 mg LY3009104, Placebo, Moxifloxacin: First Intervention: 40-mg LY3009104 dose administered orally once.
  Second Intervention: Placebo tablets (matching 40-mg LY3009104) administered orally once.
  Third Intervention: A single 400-mg moxifloxacin tablet administered orally once.
  There was a washout of at least 3 days between each intervention.
- Part B: Placebo, Moxifloxacin, 40 mg LY3009104: First Intervention: Placebo tablets (matching 40-mg LY3009104) administered orally once.
  Second Intervention: A single 400-mg moxifloxacin tablet administered orally once.
  Third Intervention: 40-mg LY3009104 dose administered orally once.
  There was a washout of at least 3 days between each intervention.
- Part B: Moxifloxacin, 40 mg LY3009104, Placebo: First Intervention: A single 400-mg moxifloxacin tablet administered orally once.
  Second Intervention: 40-mg LY3009104 dose administered orally once.
  Third Intervention: Placebo tablets (matching 40-mg LY3009104) administered orally once.
  There was a washout of at least 3 days between each intervention.
- Part B: Moxifloxacin, Placebo, 40 mg LY3009104: First Intervention: A single 400-mg moxifloxacin tablet administered orally once.
  Second Intervention: Placebo tablets (matching 40-mg LY3009104) administered orally once.
  Third Intervention: 40-mg LY3009104 dose administered orally once.
  There was a washout of at least 3 days between each intervention.
- Part B: 40 mg LY3009104, Moxifloxacin, Placebo: First Intervention: 40-mg LY3009104 dose administered orally once.
  Second Intervention: A single 400-mg moxifloxacin tablet administered orally once.
  Third Intervention: Placebo tablets (matching 40-mg LY3009104) administered orally once.
  There was a washout of at least 3 days between each intervention.
- Part B: Placebo, 40 mg LY3009104, Moxifloxacin: First Intervention: Placebo tablets (matching 40-mg LY3009104) administered orally once.
  Second Intervention: 40-mg LY3009104 dose administered orally once.
  Third Intervention: A single 400-mg moxifloxacin tablet administered orally once.
  There was a washout of at least 3 days between each intervention.
Period: First Intervention and Washout Period 1
Arm/Group | Part A: Placebo, 30 mg LY3009104, 40 mg LY3009104 | Part A: 20 mg LY3009104, 30 mg LY3009104, Placebo | Part A: 20 mg LY3009104, Placebo, 40 mg LY3009104 | Part B: 40 mg LY3009104, Placebo, Moxifloxacin | Part B: Placebo, Moxifloxacin, 40 mg LY3009104 | Part B: Moxifloxacin, 40 mg LY3009104, Placebo | Part B: Moxifloxacin, Placebo, 40 mg LY3009104 | Part B: 40 mg LY3009104, Moxifloxacin, Placebo | Part B: Placebo, 40 mg LY3009104, Moxifloxacin
Started | 3 | 3 | 3 | 8 | 9 | 9 | 9 | 9 | 9
Received at Least 1 Dose of Study Drug | 3 (Across all reporting groups, study drug is LY3009104, moxifloxacin, or placebo.) | 3 | 3 | 8 | 9 | 9 | 9 | 9 | 9
Completed | 3 | 3 | 2 | 8 | 9 | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention and Washout Period 2
Arm/Group | Part A: Placebo, 30 mg LY3009104, 40 mg LY3009104 | Part A: 20 mg LY3009104, 30 mg LY3009104, Placebo | Part A: 20 mg LY3009104, Placebo, 40 mg LY3009104 | Part B: 40 mg LY3009104, Placebo, Moxifloxacin | Part B: Placebo, Moxifloxacin, 40 mg LY3009104 | Part B: Moxifloxacin, 40 mg LY3009104, Placebo | Part B: Moxifloxacin, Placebo, 40 mg LY3009104 | Part B: 40 mg LY3009104, Moxifloxacin, Placebo | Part B: Placebo, 40 mg LY3009104, Moxifloxacin
Started | 3 | 3 | 2 | 8 | 9 | 9 | 9 | 9 | 9
Completed | 3 | 3 | 2 | 8 | 9 | 9 | 9 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Third Intervention
Arm/Group | Part A: Placebo, 30 mg LY3009104, 40 mg LY3009104 | Part A: 20 mg LY3009104, 30 mg LY3009104, Placebo | Part A: 20 mg LY3009104, Placebo, 40 mg LY3009104 | Part B: 40 mg LY3009104, Placebo, Moxifloxacin | Part B: Placebo, Moxifloxacin, 40 mg LY3009104 | Part B: Moxifloxacin, 40 mg LY3009104, Placebo | Part B: Moxifloxacin, Placebo, 40 mg LY3009104 | Part B: 40 mg LY3009104, Moxifloxacin, Placebo | Part B: Placebo, 40 mg LY3009104, Moxifloxacin
Started | 3 | 3 | 2 | 8 | 9 | 9 | 9 | 8 | 9
Completed | 3 | 3 | 2 | 8 | 9 | 9 | 9 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of LY3009104, moxifloxacin, or placebo and had at least 1 postdose safety assessment.
Groups:
- Part A (LY3009104 or Placebo): Participants were randomized to 1 of 3 treatment sequences during Part A of the study and received a single dose (LY3009104 or placebo) in each period separated by a washout of at least 3 days. LY3009104 was administered as either 20-milligrams (mg), 30-mg or 40-mg dose.
- Part B (LY3009104, Moxifloxacin, or Placebo): Participants were randomized to 1 of 6 treatment sequences during Part B of the study and received a single dose (LY3009104, moxifloxacin, or placebo) in each period separated by a washout of at least 3 days. LY3009104 was administered as a 40-mg dose. Moxifloxacin was administered as a 400-mg tablet.
- Total: Total of all reporting groups
Arm/Group | Part A (LY3009104 or Placebo) | Part B (LY3009104, Moxifloxacin, or Placebo) | Total
Number analyzed (Participants) | 9 | 53 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (15.4) | 39.9 (11.3) | 40.8 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 5 | 43 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 21 | 24
  Not Hispanic or Latino | 6 | 32 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 12 | 13
  White | 8 | 39 | 47
  More than 1 race | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 53 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Through 24 Hours Postdose in Population-Corrected QT (QTcP) Interval
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and is calculated from electrocardiogram (ECG) data. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between 2 R waves. Using the population-corrected formula: QTcP = QT/RR^beta, where beta is the population correction factor computed from a log-linear model (ln) QT = alpha+beta*ln RR fitted to all Day -1 and Day 1 predose QT and RR measurements in all periods for all participants. Baseline is the average of data collected for 2 hours before dosing on Day 1 of each period [-2 hours (h), -1.5 h, -1 h, -0.5 h, and 0 h]. The QTcP interval was not assessed during Part A of the study, as specified in the protocol. The QTcP interval at 1 h, 2 h, and 4 h postdose for moxifloxacin was compared to placebo to establish assay sensitivity.
Time Frame: Part B, Periods 1 through 3: Baseline, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 12 h, and 24 h postdose
Population: Participants enrolled in Part B of the study who had at least 1 dose of study drug (LY3009104, moxifloxacin, or placebo).
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Groups:
- Part B: Placebo: Placebo tablets (matching LY3009104) administered orally once in any period during Part B of the study.
- Part B: 40 mg LY3009104: A 40-milligram (mg) dose of LY3009104 administered orally once in any period during Part B of the study.
- Part B: Moxifloxacin: A single 400-mg moxifloxacin tablet administered orally once in any period during Part B of the study.
Arm/Group | Part B: Placebo | Part B: 40 mg LY3009104 | Part B: Moxifloxacin
Number analyzed (Participants) | 52 | 53 | 53
milliseconds (msec)
  1 h postdose (n=52, 53, 53) | -2.5 (4.9) | -2.4 (5.0) | 9.7 (5.8)
  1.5 h postdose (n=52, 53, 53) | -1.7 (3.9) | 0.1 (5.5) | 9.3 (5.8)
  2 h postdose (n=52, 53, 53) | -1.4 (6.5) | -0.1 (5.3) | 9.5 (6.9)
  3 h postdose (n=52, 53, 53) | -2.8 (5.7) | -2.5 (4.9) | 9.2 (6.2)
  4 h postdose (n=52, 53, 53) | -1.3 (5.2) | -0.8 (6.2) | 9.9 (5.5)
  6 h postdose (n=51, 53, 53) | -1.3 (8.3) | -2.2 (8.1) | 5.5 (7.3)
  12 h postdose (n=52, 52, 52) | -1.0 (8.3) | 0.8 (6.6) | 5.9 (7.6)
  24 h postdose (n=52, 53, 53) | -1.6 (6.1) | -0.8 (6.7) | 3.4 (5.5)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: 40 mg LY3009104; Test type: Superiority or Other; Least squares (LS) mean difference = 0.239, 90% CI 2-sided [-1.65 to 2.12] — LS mean difference (LY3009104 minus placebo) of change in QTcP 1 h postdose analyzed using analysis of covariance (ANCOVA) model adjusted for baseline QTc, treatment, time, period, sequence, treatment-by-time, participant, and participant-by-period
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: 40 mg LY3009104; Test type: Superiority or Other; LS mean difference = 1.81, 90% CI 2-sided [-0.0790 to 3.69] — LS mean difference (LY3009104 minus placebo) of change in QTcP at 1.5 h postdose was analyzed using an ANCOVA model adjusted for baseline QTc, treatment, time, period, sequence, treatment-by-time, participant, and participant-by-period
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: 40 mg LY3009104; Test type: Superiority or Other; LS Mean Difference = 1.44, 90% CI 2-sided [-0.446 to 3.32] — LS mean difference (LY3009104 minus placebo) of change in QTcP at 2 h postdose was analyzed using an ANCOVA model adjusted for baseline QTc, treatment, time, period, sequence, treatment-by-time, participant, and participant-by-period
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: 40 mg LY3009104; Test type: Superiority or Other; LS mean difference = 0.468, 90% CI 2-sided [-1.42 to 2.35] — LS mean difference (LY3009104 minus placebo) of change in QTcP at 3 h postdose was analyzed using an ANCOVA model adjusted for baseline QTc, treatment, time, period, sequence, treatment-by-time, participant, and participant-by-period
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: 40 mg LY3009104; Test type: Superiority or Other; LS mean difference = 0.702, 90% CI 2-sided [-1.18 to 2.59] — LS mean difference (LY3009104 minus placebo) of change in QTcP at 4 h postdose was analyzed using an ANCOVA model adjusted for baseline QTc, treatment, time, period, sequence, treatment-by-time, participant, and participant-by-period
Statistical Analysis 6: Comparison: Part B: Placebo vs Part B: 40 mg LY3009104; Test type: Superiority or Other; LS mean difference = -0.788, 90% CI 2-sided [-2.68 to 1.10] — LS mean difference (LY3009104 minus placebo) of change in QTcP at 6 h postdose was analyzed using an ANCOVA model adjusted for baseline QTc, treatment, time, period, sequence, treatment-by-time, participant, and participant-by-period
Statistical Analysis 7: Comparison: Part B: Placebo vs Part B: 40 mg LY3009104; Test type: Superiority or Other; LS mean difference = 1.71, 90% CI 2-sided [-0.182 to 3.60] — LS mean difference (LY3009104 minus placebo) of change in QTcP at 12 h postdose was analyzed using an ANCOVA model adjusted for baseline QTc, treatment, time, period, sequence, treatment-by-time, participant, and participant-by-period
Statistical Analysis 8: Comparison: Part B: Placebo vs Part B: 40 mg LY3009104; Test type: Superiority or Other; LS mean difference = 0.963, 90% CI 2-sided [-0.921 to 2.85] — LS mean difference (LY3009104 minus placebo) of change in QTcP at 24 h postdose was analyzed using an ANCOVA model adjusted for baseline QTc, treatment, time, period, sequence, treatment-by-time, participant, and participant-by-period
Statistical Analysis 9: Comparison: Part B: Placebo vs Part B: Moxifloxacin; Test type: Superiority or Other; LS mean difference = 12.3, 90% CI 2-sided [10.0 to 14.5] — LS mean difference (moxifloxacin minus placebo) of change in QTcP at 1 h postdose was analyzed using an ANCOVA model adjusted for baseline QTc, treatment, time, period, sequence, treatment-by-time, participant, and participant-by-period
Statistical Analysis 10: Comparison: Part B: Placebo vs Part B: Moxifloxacin; Test type: Superiority or Other; LS mean difference = 11.0, 90% CI 2-sided [8.74 to 13.3] — LS mean difference (moxifloxacin minus placebo) of change in QTcP at 2 h postdose was analyzed using an ANCOVA model adjusted for baseline QTc, treatment, time, period, sequence, treatment-by-time, participant, and participant-by-period
Statistical Analysis 11: Comparison: Part B: Placebo vs Part B: Moxifloxacin; Test type: Superiority or Other; LS mean difference = 11.1, 90% CI 2-sided [8.87 to 13.4] — LS mean difference (moxifloxacin minus placebo) of change in QTcP at 4 h postdose was analyzed using an ANCOVA model adjusted for baseline QTc, treatment, time, period, sequence, treatment-by-time, participant, and participant-by-period

2. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3009104
Time Frame: Parts A and B, Periods 1 through 3: Predose and 0.5 hours (h), 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 12 h, 24 h, 36 h, 48 h after administration of study drug
Population: Randomized participants who received at least 1 dose of LY3009104.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per liter (nmol/L)
Groups:
- Part A: 20 mg LY3009104: A 20-milligram (mg) LY3009104 dose administered orally once in Part A, Period 1 of the study.
- Part A: 30 mg LY3009104: A 30-mg LY3009104 dose administered orally once in Part A, Period 2 of the study.
- Part A: 40 mg LY3009104: A 40-mg LY3009104 dose administered orally once in Part A, Period 3 of the study.
- Part B: 40 mg LY3009104: A 40-mg LY3009104 dose administered orally once in any period during Part B of the study.
Arm/Group | Part A: 20 mg LY3009104 | Part A: 30 mg LY3009104 | Part A: 40 mg LY3009104 | Part B: 40 mg LY3009104
Number analyzed (Participants) | 6 | 6 | 5 | 53
nanomoles per liter (nmol/L) | 578 (28) | 734 (14) | 1270 (13) | 741 (33)

3. Primary Outcome: Pharmacokinetics: Area Under the Concentration Curve From Time 0 to Infinity [AUC(0-inf)] of LY3009104
Time Frame: as for outcome 2
Population: Randomized participants who received at least 1 dose of LY3009104 and had a predose and at least 1 postdose blood draw for AUC assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomoles per liter (h*nmol/L)
Arm/Group | Part A: 20 mg LY3009104 | Part A: 30 mg LY3009104 | Part A: 40 mg LY3009104 | Part B: 40 mg LY3009104
Number analyzed (Participants) | 5 | 6 | 5 | 53
hours*nanomoles per liter (h*nmol/L) | 3960 (27) | 5480 (19) | 8490 (14) | 6440 (26)

4. Primary Outcome: Number of Participants With 1 or More Drug-Related Adverse Events (AEs) or Any Serious AEs (SAEs)
Description: The number of participants with treatment-emergent adverse events (TEAEs) or treatment-emergent SAEs considered by the investigator to be related to study drug is reported. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through study completion and 30-day follow-up
Population: Enrolled participants who had at least 1 dose of study drug (LY3009104, moxifloxacin, or placebo) during the study.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Placebo: Placebo tablets [matching 20-milligrams (mg), 30-mg, or 40-mg LY3009104] administered orally once in any period during Part A of the study.
- Part A: 20 mg LY3009104: A 20-mg LY3009104 dose administered orally once in Part A, Period 1 of the study.
- Part B: Placebo: Placebo tablets (matching 40-mg LY3009104) administered orally once in any period during Part B of the study.
Arm/Group | Part A: Placebo | Part A: 20 mg LY3009104 | Part A: 30 mg LY3009104 | Part A: 40 mg LY3009104 | Part B: Placebo | Part B: 40 mg LY3009104 | Part B: Moxifloxacin
Number analyzed (Participants) | 8 | 6 | 6 | 5 | 52 | 53 | 53
Participants
  Drug-Related TEAE | 0 | 0 | 1 | 0 | 5 | 5 | 5
  Drug-Related SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Part A: Placebo | Part A: 20 mg LY3009104 | Part A: 30 mg LY3009104 | Part A: 40 mg LY3009104 | Part B: Placebo | Part B: 40 mg LY3009104 | Part B: Moxifloxacin
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/5 | 0/52 | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 2/8 | 1/6 | 2/6 | 0/5 | 8/52 | 6/53 | 7/53
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=8) | Part A: 20 mg LY3009104 (N=6) | Part A: 30 mg LY3009104 (N=6) | Part A: 40 mg LY3009104 (N=5) | Part B: Placebo (N=52) | Part B: 40 mg LY3009104 (N=53) | Part B: Moxifloxacin (N=53)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days